CLINICAL TRIAL: NCT03316352
Title: Ultrasound-assisted Versus Conventional Landmark-guided Paramedian Spinal Anesthesia in Elderly Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Associate professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1708-113-879
Record Dates: First submitted 2017-10-16; First posted 2017-10-20 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Anesthesia, Spinal; Ultrasonography
MeSH Terms: interventions — Congresses as Topic; Ultrasonography; Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound-assisted (Experimental): Ultrasound-assisted paramedian technique spinal anesthesia will be performed. A Preprocedural ultrasound scan will be performed for skin marking of entry site of spinal needle. Spinal anesthesia will be performed via paramedian approach using the skin marking site as entry point. 0.5% heavy bupivacaine will be administered into intrathecal space.
  Interventions: Procedure: Ultrasound-assisted paramedian technique spinal anesthesia; Device: Ultrasound; Drug: 0.5% heavy bupivacaine
- Landmark-guided (Active Comparator): In these patients, spinal anesthesia will be performed via paramedian approach using conventional landmark palpation technique. Landmark-guided paramedian technique spinal anesthesia will be performed. 0.5% heavy bupivacaine will be administered into intrathecal space.
  Interventions: Procedure: Landmark-guided paramedian technique spinal anesthesia; Drug: 0.5% heavy bupivacaine

INTERVENTIONS:
Procedure: Ultrasound-assisted paramedian technique spinal anesthesia — Ultrasound-assisted paramedian technique will be used. A preprocedural ultrasound scan will be performed, and skin marking for spinal entry site will be done using ultrasound scan. Spinal anesthesia will be done according to skin marking using ultrasound, via paramedian approach.
  Other Names: sono-assisted
  Arms: Ultrasound-assisted
Procedure: Landmark-guided paramedian technique spinal anesthesia — Landmark-guided paramedian technique will be used. Spinal anesthesia will be done using conventional landmark-guided paramedian technique.
  Other Names: conventional
  Arms: Landmark-guided
Device: Ultrasound — A preprocedural ultrasound scan will be done using Portable Echocardiography system (Vivid-i, GE healthcare) with 4C-RS convex probe (2.0-5.5 MHz Frequency range).
  Other Names: sonography
  Arms: Ultrasound-assisted
Drug: 0.5% heavy bupivacaine — During spinal anesthesia, 0.5% heavy bupivacaine will be administered into intrathecal space. The dose of local anesthetic injected for spinal anesthesia will be at the discretion of the attending anesthesiologist. The dose range of intrathecal bupivacaine will be between 12 and 16 mg.
  Other Names: bupivacaine

SUMMARY:
Multiple passes and attempts during spinal anesthesia might be associated with a greater incidence of paraesthesia, postdural puncture headache, and spinal hematoma. We hypothesized that the use of a preprocedural ultrasound-assisted paramedian technique for spinal anesthesia in patients with old age would reduce the number of passes required to entry into the subarachnoid space when compared with the landmark-guided paramedian approach. The study participants will be randomized into group L (landmark-guided) and group U (ultrasound-assisted). In group L, spinal anesthesia will be performed via paramedian approach using conventional landmark palpation technique. In group U, a preprocedural ultrasound scan will be used to mark the needle insertion site, and spinal anesthetic will be done via the paramedian approach.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients (age≥60 years) scheduled to undergoing elective orthopedic surgery under spinal anesthesia
* Patients with ASA physical status classification I, II, III

Exclusion Criteria:

* Patients with contraindication to spinal anesthesia (coagulopathy, local infection, allergy to local anesthetic)
* Patients with morbid cardiac diseases
* Pregnancy
* Patients with previous history of lumbar spine surgery

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2018-01-11 (Actual); Study Completion 2018-01-11 (Actual)

PRIMARY OUTCOMES:
the number of needle passes | from the initiation of spinal anesthesia procedure, until the completion of spinal anesthetic injection
  the number of forward advancements of the spinal needle in a given interspinous space, i.e., withdrawal and redirection of spinal needle without exiting the skin

SECONDARY OUTCOMES:
Number of spinal needle insertion attempts | from the initiation of spinal anesthesia procedure, until the completion of spinal anesthetic injection
  the number of times the spinal needle was withdrawn from the skin and reinserted
Time for identifying landmarks | from the initiation of spinal anesthesia procedure, until the completion of spinal anesthetic injection
  In group L, time from start of palpation to completion of the process, as declared by the anesthesiologist. In group U, time from placement of the ultrasound probe on the skin to the completion of markings.
Time taken for performing spinal anesthetic | from the initiation of spinal anesthesia procedure, until the completion of spinal anesthetic injection
  time from needle insertion to the completion of injection
Level of block | 5, 10, 15 minutes after the completion of spinal anesthetic injection
  loss of cold sensation tested with 2% chlorhexidine swab
Incidence of radicular pain, paraesthesia, and blood tapping in the spinal needle | from the initiation of spinal anesthesia procedure, until the completion of spinal anesthetic injection
  Incidence of radicular pain, paraesthesia, and blood tapping in the spinal needle during the spinal anesthesia procedure
Periprocedural pain | from the initiation of spinal anesthesia procedure, until the completion of spinal anesthetic injection
  11-point verbal rating scale (0=no pain, 10=most pain imaginable)
Periprocedural discomfort score | from the initiation of spinal anesthesia procedure, until the completion of spinal anesthetic injection
  11-point verbal rating scale (0=no discomfort, 10=most discomfort imaginable)

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kallidaikurichi Srinivasan K, Iohom G, Loughnane F, Lee PJ. Conventional Landmark-Guided Midline Versus Preprocedure Ultrasound-Guided Paramedian Techniques in Spinal Anesthesia. Anesth Analg. 2015 Oct;121(4):1089-1096. doi: 10.1213/ANE.0000000000000911. PMID 26270115
- [Background] Chin KJ, Perlas A, Chan V, Brown-Shreves D, Koshkin A, Vaishnav V. Ultrasound imaging facilitates spinal anesthesia in adults with difficult surface anatomic landmarks. Anesthesiology. 2011 Jul;115(1):94-101. doi: 10.1097/ALN.0b013e31821a8ad4. PMID 21572316
- [Derived] Park SK, Yoo S, Kim WH, Lim YJ, Bahk JH, Kim JT. Ultrasound-assisted vs. landmark-guided paramedian spinal anaesthesia in the elderly: A randomised controlled trial. Eur J Anaesthesiol. 2019 Oct;36(10):763-771. doi: 10.1097/EJA.0000000000001029. PMID 31188153